CLINICAL TRIAL: NCT03013634
Title: Protective Effects of Dexmedetomidine on Myocardial Injury During Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin First Central Hospital (Other)
Responsible Party: Principal Investigator, Wenli Yu, Wenli Yu,PhD ,Department of Anesthesiology,Tianjin First Center Hospital, Tianjin First Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TianjinFCH
Record Dates: First submitted 2016-12-22; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Evidence of Liver Transplantation; Myocardial Injury
Keywords: dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine Group (Experimental): Dexmedetomidine infusion:loading 0.5ug/kg for 10min, then 0.5 ug/kg/h until the end of operation.
  Interventions: Drug: Dexmedetomidine
- Normal saline Group (Placebo Comparator): Equal volume normal saline substitute for dexmedetomidine
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine infusion:loading 0.5ug/kg for 10min, then 0.5 ug/kg/h until the end of operation.
  Arms: Dexmedetomidine Group
Drug: Normal saline — Equal volume normal saline substitute for dexmedetomidine
  Arms: Normal saline Group

SUMMARY:
The purpose of this study was to evaluate the protective effect of dexmedetomidine on myocardial injury during liver transplantation

DETAILED DESCRIPTION:
Liver transplantation surgery may lead to myocardial injury. Dexmedetomidine, a highly specific α2-adrenoeptor agonist, has sedative and analgesic properties without significant respiratory depression at the clinically approved dosage. Some investigations indicated that dexmedetomidine was able to protect the myocardium via improving the activity of Na+-K+-adenosine triphosphate enzyme and Ca2+-adenosine triphosphate, alleviating inflammation reaction and avoiding Ca2+ overload. However, the effect and the mechanism of dexmedetomidine on myocardial injury during liver transplantation remain unclear.

ELIGIBILITY:
Inclusion Criteria:

* End stage liver disease scheduled for liver transplantation in Tianjin First Center Hospital

Exclusion Criteria:

* Pre-existing respiratory failure,renal failure,hepatic encephalopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Peri-operative mortality | through study completion, an average of 5 weeks
The incidence of cardiac complications | from anesthesia induction to 24 hours after operation

SECONDARY OUTCOMES:
Evidences of Clinically Definite Myocardial Injury Confirmed by Electrochemiluminescence | before skin incision, 0.5 hour min after anhepatic, 2 hours of neohepatic stage,the end of surgery,24 hours after operation
  myohemoglobin,creatine kinase isoenzyme,cardiac troponinⅠ,Heart-type fatty acid-binding protein

OTHER OUTCOMES:
Length of ICU stay | through study completion, an average of 5 days
length of stay | through study completion, an average of 6 weeks
  from date of admission to discharge time

CONTACTS AND LOCATIONS:
Locations (1):
- No.24 Fukang Road,Nankai District, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No